CLINICAL TRIAL: NCT06651580
Title: Pediatric Longitudinal Cohort Study of Chronic Pancreatitis (INSPPIRE 2)
Brief Title: Biospecimen Collection to Identify Gene Mutations for High Risk Pancreatic Cancer in Pediatric Patients, INSPPIRE 2 Study
Status: Recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2020-1057; NCI-2021-04028 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-1057 (Other: M D Anderson Cancer Center); P30CA016672 (NIH)
Record Dates: First submitted 2024-10-18; First posted 2024-10-21 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Chronic Pancreatitis; Exocrine Pancreas Carcinoma; Recurrent Acute Pancreatitis
MeSH Terms: conditions — Pancreatitis, Chronic; Pancreatic Neoplasms; Pancreatitis | interventions — Specimen Handling

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, saliva, urine, or stool samples

GROUPS / COHORTS (1):
- Observational (biospecimen collection and questionnaire): Patients complete QoL assessment and complete questionnaires for over 2 hours every 12 months for 4 years. Patients also undergo collection of blood and/or saliva (if blood samples are not available), urine, or stool at baseline.
  Interventions: Procedure: Biospecimen Collection; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood, saliva, urine or stool samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Other: Quality-of-Life Assessment — Complete QoL assessment
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Complete questionnaire

SUMMARY:
This clinical trial collects blood, saliva, urine, or stool samples to help identify possible genetic mutations that may increase a person's chance at developing pancreatic cancer. Finding genetic markers among pediatric patients with acute recurrent pancreatitis and chronic pancreatitis may help identify patients who are at risk of pancreatic cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To comprehensively characterize the pediatric population with acute recurrent pancreatitis (ARP) and chronic pancreatitis (CP) and determine predictors of early onset CP and its sequelae.

OUTLINE:

Patients complete quality-of-life (QoL) assessment and complete questionnaires for over 2 hours every 12 months for 4 years. Patients also undergo collection of blood and/or saliva (if blood samples are not available), urine, or stool at baseline or follow-up (if inadequate samples collected or missed at baseline).

After completion of the study, patients are followed up every 12 months.

ELIGIBILITY:
Inclusion Criteria:

* All subjects/parents must sign an informed consent and/or assent indicating that they are aware of the investigational nature of this study
* Subjects/parents must have signed an authorization for the release of their or their child's protected health information
* All children must be under 18 years of age at the time of enrollment
* All children providing samples should fit the ARP or CP inclusion criteria defined below:

  * Acute pancreatitis (AP): AP is defined as requiring 2 of the following:

    * Abdominal pain compatible with AP
    * Serum amylase and/or lipase values >= 3 times upper limits of normal
    * Imaging findings of AP, such as gland enlargement, acute inflammatory changes, and fluid collections
  * ARP is defined as: At least 2 episodes of acute pancreatitis with complete resolution of pain and a >= 1 month pain-free interval between episodes
  * Chronic Pancreatitis:

    * Children with at least:

      * One irreversible structural change in the pancreas with or without abdominal pain +/- exocrine pancreatic insufficiency +/- diabetes

        * Irreversible structural changes:

          * Ductal calculi, dilated side branches, parenchymal calcifications found in any imaging (abdominal ultrasound [abd US], magnetic resonance imaging/magnetic resonance cholangiopancreatography [MRI/MRCP], computerized tomography [CT], endoscopic retrograde cholangiopancreatography [ERCP], endoscopic US [EUS])
          * Ductal obstruction or stricture/dilatation/irregularities that are persistent (for >= 2 months) on any imaging
          * Parenchymal atrophy, irregular contour, accentuated lobular architecture, cavities alone are not diagnostic findings for CP
          * Surgical or pancreatic biopsy specimen demonstrating histopathologic features compatible with CP (acinar atrophy, fibrosis, protein plugs, infiltration with lymphocytes, plasma cells, macrophages)

Exclusion Criteria:

* Subjects must not have any significant medical illnesses that in the investigator's opinion cannot be adequately controlled with appropriate therapy or would compromise the subject's ability to tolerate study interventions

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric patients (under 18 years) enrolled in the INSPPIRE 1 database who are planned to be reenrolled under this protocol over the next 4 years.
Sampling Method: Non-Probability Sample
Enrollment: 1600 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2027-02-02 (Estimated); Study Completion 2027-02-02 (Estimated)

PRIMARY OUTCOMES:
Characterize the pediatric population with acute recurrent pancreatitis (ARP) and chronic pancreatitis (CP) | Up to 4 years
  Two-sample t-test or Wilcoxon rank-sum test will be used for the continuous/ordinal variables and Pearson Chi-square test for the categorical variables. The variables that suggest differences between ARP and CP (p value < 0.15) will be included as independent variables in a multivariable logistic regression analysis for CP progression.
Risk factors that predispose children to CP sequelae and high disease burden | Up to 4 years
  A two-sample t-test or Wilcoxon rank-sum test for the continuous/ordinal variables and Pearson Chi-square test for the categorical variables. The variables that suggest an association with sequelae/disease burden (p-value < 0.15) will be included as independent variables in a regression model for sequelae/disease burden. Normal/logistic/multinomial regression model will be used for continuous/binary/ordinal disease burden and sequelae outcomes. For repeated measures, random effects will be added to these models to account for correlation among the measures.

CONTACTS AND LOCATIONS:
Overall Officials: Ying Yuan, PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (26):
- United States (22):
  - Children's Hospital Los Angeles, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - University of Colorado, Denver, Colorado
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Riley Hospital for Children, Indianapolis, Indiana
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Boston Children's Hospital, Boston, Massachusetts
  - University of Minnesota/Masonic Children's Hospital, Minneapolis, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - University of Texas Southwestern/Children's Medical Center, Dallas, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Texas Children's Hospital, Houston, Texas
  - Children's Hospital of San Antonio, San Antonio, Texas
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Sydney Children's Hospital, Randwick, New South Wales, Australia
- Canada (2):
  - Hospital for Sick Children, Toronto, Ontario
  - The Montreal Children's Hospital of the MUHC, Montreal, Quebec
- Hadassah University Hospital, Jerusalem, Israel